CLINICAL TRIAL: NCT06816277
Title: Application of Local Melatonin for Controlling Peri-implant Diseases: a Randomized Clinical Trial
Brief Title: Application of Local Melatonin in Peri-implantitis
Acronym: MEL19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C.I. 19/313-E; 2019-000828-18 (EudraCT Number)
Record Dates: First submitted 2025-01-07; First posted 2025-02-10 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Periimplantitis
Keywords: melatonin; periimplant disease; marginal bone loss; inflammation; treatment
MeSH Terms: conditions — Peri-Implantitis; Inflammation

STUDY DESIGN:
Intervention Model Description: Two blinded groups
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Letter and number code randomized assigned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonina (Experimental): El tratamiento periimplantario y el desbridamiento mecánico se realizarán en todos los casos bajo anestesia local convencional. El procedimiento seguirá la secuencia habitual en todos los casos. El acceso quirúrgico se hará a través de una incisión intrasulcular y lineal, y el desprendimiento de un colgajo mucoperiostéico. El tratamiento peri-implante se realizará con una punta de ultrasonido bajo irrigación, complementada con el uso de curetas si es necesario. Posteriormente, en los casos del grupo correspondiente, se aplicará melatonina (1,9 mg) a la cama periimplantacional. Suturado con seda monofilamento 4/0 en una aguja semicircular de 3/8 premontada. Después de 7 días, se revisará el proceso de curación y se eliminarán las suturas.
  Interventions: Procedure: Desbridamiento de periimplantitis; Drug: Aplicación de melatonina; Other: Placebo application
- Placebo (Placebo Comparator): The peri-implant treatment and mechanical debridement will be performed in all cases under conventional local anesthesia. The procedure will follow the usual sequence in all cases. Surgical access will be made through an intrasulcular and linear incision, and the detachment of a mucoperiosteal flap. The peri-implant treatment will be performed with an ultrasound tip under irrigation, complemented by the use of curettes if necessary. Subsequently, in the cases of the corresponding group, melatonin (1.9 mg) will be applied to the peri-implant bed.
  sutured with 4/0 monofilament silk on a pre-mounted 3/8 semicircular needle. After 7 days, the healing process will be reviewed and the sutures will be removed.
  Interventions: Procedure: Desbridamiento de periimplantitis; Drug: Aplicación de melatonina; Other: Placebo application

INTERVENTIONS:
Procedure: Desbridamiento de periimplantitis — The implant with the most severe involvement was selected, although the treatment was performed on all implants, to prevent patients with more affected implants from having greater statistical relevance.
  The peri-implant surgical treatment was performed under local infiltrative anesthesia with 4% articaine with 1:100,000 adrenaline. Debridement was performed using ultrasound with irrigation, complemented using curettes. Treatment with melatonin or placebo was applied through computer block randomization. To achieve blinding, a different code was assigned to the group applying 1.9 mg of melatonin (A) and to the control group (B) applying placebo (dextrinomaltose 2 mg) powder and the samples and records were coded. It was sutured with 4/0 monofilament in a pre-assembled 3/8 s
Drug: Aplicación de melatonina — Treatment with melatonin or placebo was applied through computer block randomization. To achieve blinding, a different code was assigned to the group applying 1.9 mg of melatonin (A) and to the control group (B) applying placebo (dextrinomaltose 2 mg) powder and the samples and records were coded.
Other: Placebo application — Treatment with melatonin or placebo was applied through computer block randomization. To achieve blinding, a different code was assigned to the group applying 1.9 mg of melatonin (A) and to the control group (B) applying placebo (dextrinomaltose 2 mg) powder and the samples and records were coded.

SUMMARY:
A randomized clinical trial was carried out in patients affected by peri-implantitis with a follow-up of 60 days. Melatonin 1.9 mg or placebo was applied locally to the peri-implant defect after nonsurgical debridement.

To determine the effectiveness anti-inflammatory, osteogenic and antimicrobial properties were evaluated. The probing depth, bleeding index, plaque index, and interleukin-1β and 6 concentrations, peri-implant bone level and the bacterial strains were analyzed.

DETAILED DESCRIPTION:
This randomized clinical trial was conducted following the recommendations of the Consolidated Standards of Reporting Trials Statement (CONSORT 2010), the requirements set out in the Declaration of Helsinki (World Medical Assembly) and in accordance with the Data Protection Law (Organic Law 3/2018, of December 5, on the Protection of Personal Data and the guarantee of digital rights). The protocol was approved by the Clinical Research Ethics Committee (CEIC) of the Hospital Clínico San Carlos de Madrid, minute 7.2/19; C.P. MEL19 - C.I. 19/313-E. In Spain, the Spanish Agency for Medicines and Health Products (AEMPS), dependent on the Ministry of Health, establishes that the use of melatonin in doses higher than 1.9 mg was only possible under medical prescription for the treatment of sleep disorders and hyperactivity disorders, or autism spectrum (Royal Legislative Decree 1/2015), which is why it is only marketed in Spain in doses lower than 2 mg. Recruitment Volunteer participants diagnosed with peri-implant disease were recruited according to the criteria of the Classification of Periodontal and Peri-implant Diseases and Conditions of the 2017 Global Workshop, with an indication for peri-implant surgical treatment, with one or more fully erupted teeth.

Patients of both sexes, aged between 40 and 85 years, in good health (Category I and II of the American Society of Anesthesiologists [ASA]), with no history or metabolic or systemic diseases affecting the bone or the healing process, such as diabetes, without autoimmune diseases, autoimmune coagulation or healing disorders and who, meeting the inclusion criteria, agreed to sign the informed consent were included. Exclusion criteria were established as tobacco consumption >25 cigarettes per day, the use of hormones, anti-inflammatories, corticosteroids, immunosuppressants, analgesics, antidiabetic or antiresorptive medications regularly or recently, pregnant or lactating women, and those who refused to participate in the study or did not allow follow-up and sample collection. Study design: The most severely affected implant was selected, although treatment was performed on all implants, to avoid patients with more severely affected implants having a greater statistical significance. Before treatment (T0), the peri-implant clinical and radiological study was carried out using periapical radiography with a parallelism and crevicular fluid samples were obtained from the implant in duplicate. Peri-implant surgical treatment was performed under local infiltration anesthesia with 4% articaine with 11,000,000 adrenaline. Debridement was performed using ultrasound with irrigation, supplemented with curettes.

Melatonin or placebo treatment was applied through computer block randomization. To achieve blinding, a different code was assigned to the group that applied 1.9 mg of melatonin (A) and the control group (B) that applied placebo powder (dextrinomaltose 2 mg) and the samples and records were coded. It was sutured with 4/0 monofilament on a pre-mounted 3/8 semicircular needle. In all patients, 1000 mg of paracetamol was prescribed every 8 hours in case of pain, and they were instructed not to rinse or use any topical antiseptic. At 7 days (T1), the healing process was reviewed, the sutures were removed and crevicular fluid samples were taken. At 21 days (T2), a new complete peri-implant record, new crevicular fluid samples and a radiological study were performed. At 60 days (T3), a new complete peri-implant record, crevicular fluid samples and a radiological study were performed. To detect the occurrence of complications, a record of adverse events was established for a period of two months after treatment. Variables Probing depth: The distance from the gingival margin to the bottom of the periodontal pocket was considered. The measurement was carried out at the four locations surrounding the implant, mesial, distal, lingual and vestibular. In addition, the average of the four locations was presented. Plaque index (Löe and Silness) The presence of visible bacterial plaque was considered suitable for implant rehabilitation (Grade 0: No plaque; Grade 1: No plaque visible to the naked eye.

Plaque is present when probing in the peri-implant area; Grade 2: Visible bacterial plaque is present; Grade 3: Visible bacterial plaque is present surrounding the implant, including the interdental spaces. Stones may be present. Adequate plaque control is considered when the index results in a value ≤1. Bleeding index (Löe and Silness) It was considered during the 30 seconds after probing adapted to the implant model (Grade 0: No bleeding; Grade 1: A spot of blood does not appear until a few seconds after probing; Grade 2: Bleeding immediately after probing; Grade 3: Bleeding at the slightest contact with the mucosa, extension of bleeding along the sulcus). marginal bone loss Assessment of the peri-implant crestal bone level was performed using ImageJ® software (NIH, Bethesda, MD, USA). From the pixel measurement of the known implant length, the vertical bone level measurement was determined from the implant platform and perpendicular to it, to the area of the turbinate bone in contact with the implant surface both mesial and distal. It was considered as a single measurement of the mesial and distal mean of each implant taking into account the clinical importance.

IL-1β and IL-6 concentration Crevicular fluid samples obtained using Perio-paper strips were analyzed with the enzyme-linked immunosorbent assay (ELISA) technique. The samples were stored in sterile 13x75mm x 2 mL BD Vacutainer® tubes and were processed using the ELH-IL1B-1 Human IL-1 beta ELISA Kits 1 x 96-Wel BIONOVA CIENTIFICA S.L and HEA079HU-48T High Sensitive ELISA Kit for Interleukin 6 (IL-6) 48T BIONOVA CIENTIFICA SL for analysis of interleukin-1β and 6 at 60-90 minutes after obtaining it. The determinations were read using the ELISA reader (Ivymen System 2100-C). The standard curve of the kits was made in duplicate for IL-1β and IL-6 both in the test and in the total analysis of the samples.

Microbiological count: A Colon Forming Unit (CFU) count was performed on the crevicular fluid samples obtained using sterile paper points. They were transferred into a vial of reduced transport liquid with 1.0 mL of RTF transport medium to preserve the anaerobiosis of the samples for 24 hours and quantify the sample volume. The samples were immediately cultured on blood agar medium and the peri-implantopathogenic, periodontopathogenic and candida species were identified.

Sample size calculation: The calculation of the sample size was carried out taking as reference previous similar studies. 30 patients (15/15) were considered to detect differences with a large effect size (d=1) and with a statistical power of 80%. Considering a possible drop out of patients, a minimum recruitment of 33 patients was estimated.

Statistical analysis: A descriptive analysis of the most relevant statistics was carried out for all the variables collected in the research: absolute and relative frequencies (for the categorical ones) and mean, standard deviation, range, median and 25th and 75th percentiles (for the continuous ones).

The Shapiro-Wilk test was applied to evaluate the adjustment to a normal distribution of the variables in both groups. To carry out the inferential analysis, the non-parametric Brunner-Langer Model for longitudinal data was used. To study the evolution of the different variables (clinical, inflammatory, microbiological) throughout all measurements of the period depended on the type of treatment.

A level of statistical significance p≤0.05 was established.

ELIGIBILITY:
Inclusion criteria:

* Peri-implant disease was recruited according to the criteria of the 2017 World Workshop Classification of Periodontal and Peri-implant Diseases and Conditions.
* Indication for peri-implant surgical treatment.
* One or more fully erupted teeth.
* American Society of Anesthesiologists [ASA] Category I and II.
* No history or metabolic or systemic diseases affecting the bone or healing process.
* Agreed to sign informed consent.

Exclusion criteria:

* Tobacco use >25 cigarettes per day.
* Use of hormonal, anti-inflammatory, corticosteroid, immunosuppressant, analgesic, antidiabetic or antiresorptive medications on a regular or recent basis.
* Pregnant or lactating women.
* Those who refused to participate in the study or did not allow follow-up and sample collection.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Probing depth | 60 days
  The distance from the gingival margin to the bottom of the periodontal pocket was considered. The measurement was carried out in the four locations surrounding the implant, mesial, distal, lingual and vestibular. Additionally, the average of the four locations was presented.

SECONDARY OUTCOMES:
Plaque Index (Löe y Silness) | 60 days
  The presence of visible bacterial plaque was considered adapted to rehabilitation using implants (Grade 0: No plaque; Grade 1: No plaque with the naked eye. There is plaque when the exploration is performed with a probe in the peri-implant area; Grade 2: There is visible bacterial plaque; Grade 3: There is visible bacterial plaque surrounding the implant, including interdental spaces. There may be stones.
  Adequate plaque control is considered to exist when the index results in a value ≤1.
Bleeding Index (Löe y Silness) | 60 days
  It was considered during the 30 seconds after probing adapted to the implant model (Grade 0: Absence of bleeding; Grade 1: A spot of blood does not appear until a few seconds after probing; Grade 2: Bleeding immediately after of probing; Grade 3: Bleeding at the slightest contact with the mucosa, extension of bleeding along the sulcus).
Marginal bone loss | 60 days
  The evaluation of the peri-implant-crestal bone level was performed using the ImageJ® program (NIH, Bethesda, MD, USA). From the measurement in pixels of the known length of the implant, the vertical measurement of the bone level was determined from the implant platform and perpendicular to it, to the area of turbinate bone in contact with the surface of the implant both mesial and distal. It was considered as a single measurement of the mesial and distal mean of each implant considering the clinical significance .
IL-1β concentration | 60 days
  Crevicular fluid samples obtained using Perio-paper strips were analyzed with the enzyme-linked immunosorbent assay (ELISA) technique. The samples were stored in sterile 13x75mm x 2 mL BD Vacutainer® tubes and were processed using the ELH-IL1B-1 Human IL-1 beta ELISA Kits 1 x 96-Wel BIONOVA CIENTIFICA S.L and HEA079HU-48T High Sensitive ELISA Kit for Interleukin 6 (IL-6) 48T BIONOVA CIENTIFICA SL for analysis of interleukin-1β and 6 at 60-90 minutes after obtaining it. The determinations were read using the ELISA reader (Ivymen System 2100-C). The standard curve of the kits was made in duplicate for IL-1β and IL-6 both in the test and in the total analysis of the samples.
IL-6 concentration | 60 days
  Crevicular fluid samples obtained using Perio-paper strips were analyzed with the enzyme-linked immunosorbent assay (ELISA) technique. The samples were stored in sterile 13x75mm x 2 mL BD Vacutainer® tubes and were processed using the ELH-IL1B-1 Human IL-1 beta ELISA Kits 1 x 96-Wel BIONOVA CIENTIFICA S.L and HEA079HU-48T High Sensitive ELISA Kit for Interleukin 6 (IL-6) 48T BIONOVA CIENTIFICA SL for analysis of interleukin-1β and 6 at 60-90 minutes after obtaining it. The determinations were read using the ELISA reader (Ivymen System 2100-C). The standard curve of the kits was made in duplicate for IL-1β and IL-6 both in the test and in the total analysis of the samples.
Microbiological count | 60 days
  A Colon Forming Unit (CFU) count was performed on the crevicular fluid samples obtained using sterile paper points. They were transferred into a vial of reduced transport liquid with 1.0 mL of RTF transport medium to preserve the anaerobiosis of the samples for 24 hours and quantify the sample volume. The samples were immediately cultured on blood agar medium and the peri-implantopathogenic, periodontopathogenic and candida species were identified.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Specialities. Faculty of Dentistry. Complutense University of Madrid., Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
It could be shared by email to the contact person of the investigation. All data except from personal information could be available. The results will be published.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available for five years.
Access Criteria: Applicants must identify the purpose of the data request

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT06816277/Prot_SAP_ICF_000.pdf